CLINICAL TRIAL: NCT02699502
Title: Metabolic Therapy in Patients With Osteoporosis After Hip Fracture by Cooperation Orthopedic-rehabilitation-metabolic: Determination of Drug Treatment Regardless of Reaching the Follow-up Clinic
Brief Title: Metabolic Therapy in Patients With Osteoporosis After Hip Fracture by an Orthopedic-rehabilitation-metabolic Team
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0210-15-MMC
Record Dates: First submitted 2016-02-08; First posted 2016-03-04 (Estimated); Last update posted 2016-03-04 (Estimated); Status verified 2016-02

CONDITIONS: Hip Fracture
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- patients with osteoporotic hip fractures (Experimental): The intervention includes matching an appropriate drug to patients with hip fractures. All the relevant parameters regarding the patients with osteoporotic hip fractures will be reviewed (age, kidney function, previous treatment) and an appropriate anti osteoporosis medication will be determined. A recommendation regarding treatment will be sent to the local regulatory authorities, which will send the approved recommendation the the family physician.
  Interventions: Other: matching an appropriate drug therapy to patients with osteoporotic hip fractures

INTERVENTIONS:
Other: matching an appropriate drug therapy to patients with osteoporotic hip fractures — The process involves reviewing patients characteristics virtually and finding the right drug for them while they are still in the hospital. After matching an appropriate drug, getting it through regulatory authorities to the family physician

SUMMARY:
Metabolic therapy in patients with osteoporosis after hip fracture by cooperation orthopedic-rehabilitation-metabolic: Determination of drug treatment regardless of reaching the follow-up clinic

DETAILED DESCRIPTION:
Osteoporotic hip fractures are a significant cause of morbidity and mortality in older age. Patients with this fracture are at high risk of further fracture, it can be reduced by appropriate metabolic therapy. However, only 30% of patients after a hip fracture receive basic treatment appropriate calcium and vitamin D, only 10-15% receive complementary metabolic therapy more drugs prevent bone resorption, or bone-building drugs as recommended in the literature, the prevention of further fractures. studies conducted in the past have proven, multi-disciplinary team of dedicated financial institution may increase appropriate treatment and improve the quality of care in these patients.

Previous data in our institution has shown that 84% of patients with hip fractures received calcium and vitamin D during hospitalization, but only 47% of the patients came to the metabolic clinic. Moreover, of the patients who came to the metabolic clinic, only 46% were put on complementary metabolic therapy, mostly due to a lack of sufficient vitamin D level. In the present study investigators attempt to treat patients without physical attendance at the metabolic clinic.

ELIGIBILITY:
Inclusion Criteria:

* All patients were analyzed could Department of Orthopedics with a hip fracture

Exclusion Criteria:

-

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-03 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
The number of patients with hip fracture that will receive anti osteoporosis therapy without attending the metabolic clinic in comparison to previous results in the study mentioned above (No. Helsinki 0072-14-MMC) | half a year

SECONDARY OUTCOMES:
Number of drugs that will be approved by the regulatory authorities | half a year
Number of drugs that will be prescribed by family physicians | half a year

IPD SHARING:
Plan to Share IPD: No